CLINICAL TRIAL: NCT06035978
Title: Use of Determination of Drug Levels to Optimize Pharmacotherapy of Heart Failure
Brief Title: Determination of Drug Levels for Pharmacotherapy of Heart Failure
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNO-HeFa1-BESPISAVA
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Heart Failure With Reduced Ejection Fraction
Keywords: Cardiovascular Diseases; Heart Failure with Reduced Ejection Fraction
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Nebivolol; sacubitril and valsartan sodium hydrate drug combination; Carvedilol; Bisoprolol; Metoprolol; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Heart Failure with Reduced Ejection Fraction (Experimental): Patients with heart failure with reduced ejection fraction, aged 18+, dispensary at the Cardiology Outpatient Clinic for Heart Failure University Hospital Ostrava, who are orally administered tablets one of the evaluated medicinal products or their combination as indicated by the attending physician (Nebivolol, Valsartan and Sacubitril, Carvedilol, Bisoprolol, Metoprolol, Spironolactone).
  Interventions: Drug: Nebivolol; Drug: Valsartan and Sacubitril; Drug: Carvedilol; Drug: Bisoprolol; Drug: Metoprolol; Drug: Spironolactone

INTERVENTIONS:
Drug: Nebivolol — Nebivolol (Nebilet) tablet will be administered orally to patients according to their clinical condition and the decision of the attending physician.
  Other Names: Nebilet, anatomical-therapeutic-chemical code (ATC) C07AB12
Drug: Valsartan and Sacubitril — Valsartan and Sacubitril (Entresto) tablet will be administered orally to patients according to their clinical condition and the decision of the attending physician.
  Other Names: Entresto, ATC C09DX04
Drug: Carvedilol — Carvedilol (Dilatrend) tablet will be administered orally to patients according to their clinical condition and the decision of the attending physician.
  Other Names: Dilatrend, ATC C07AG02
Drug: Bisoprolol — Bisoprolol (Concor) tablet will be administered orally to patients according to their clinical condition and the decision of the attending physician.
  Other Names: Concor, ATC C07AB07
Drug: Metoprolol — Metoprolol (Betaloc ZOK) tablet will be administered orally to patients according to their clinical condition and the decision of the attending physician.
  Other Names: Betaloc ZOK, ATC C07AB02
Drug: Spironolactone — Verospiron (Spironolactone) tablet will be administered orally to patients according to their clinical condition and the decision of the attending physician.
  Other Names: Verospiron, ATC C03DA01

SUMMARY:
The aim of this study is to determine whether and how serum concentrations of the used medicinal products, including their metabolites, correlate with selected clinical indicators of heart failure (NT-proBNP concentration, 6-minute walk test, quality of life questionnaire, echocardiographic parameters, hospitalization for HFrEF, length of survival).

DETAILED DESCRIPTION:
The prevalence of chronic heart failure increases with age, and this disease is one of the most common reasons for hospitalization in the elderly. In order to reduce the number of exacerbations, the frequency of hospitalizations, morbidity and mortality and improve the overall quality of life, the treatment strategy should be individually set for each patient, regularly monitored and reviewed.

Patients with chronic heart failure show significant differences in the pharmacokinetics of both cardiovascular and non-cardiovascular drugs. At the same time, they tend to be exposed to other prescribed medicinal products, and therefore there is an increased risk of drugs interactions. These findings emphasize the need for comprehensive pharmacokinetic studies in patients with chronic heart failure, together with the exploration of the potential benefit of biomarkers suitable for monitoring the clinical status of patients. Pharmacotherapy of chronic heart failure with reduced ejection fraction (Heart Failure with Reduced Ejection Fraction - HFrEF) currently consists of beta-blockers together with mineralocorticoid receptor antagonists, the combination of sacubitril/valsartan drugs and sodium-glucose transporter 2 inhibitors. Although the recommendation of therapeutic drug monitoring (TDM) in patients with chronic heart failure has not yet been established, its introduction can serve as an effective tool for detecting changes in the pharmacokinetics of drugs used, objectifying drug interactions and ascertaining patient adherence to treatment, thereby becoming part of safe personalized pharmacotherapy of this disease.

ELIGIBILITY:
Inclusion Criteria:

* HFrEF with already established or newly started treatment with the listed medicinal products
* Male and female patients over 18 years of age
* Signed Informed Consent with participation in the study
* Women of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) result at baseline and use an acceptable method of contraception with a home control urine pregnancy test every 3 months throughout the duration of the study

Exclusion Criteria:

* Hypersensitivity to the medicinal substance or to any auxiliary substance
* Pregnant and breastfeeding women
* Additional exclusion criteria for patients taking Bisoprolol, Carvedilol, Metoprolol succinate or Nebivolol: Unstable or decompensated heart failure belonging to New York Heart Association (NYHA) group IV according to the New York Heart Association classification, requiring intravenous inotropic support
* Additional exclusion criteria for patients using Bisoprolol, Carvedilol, Metoprolol succinate or Nebivolol:
* - Clinically manifest liver dysfunction
* - History of bronchospasm or asthma
* - Severe obstructive airways disease
* - 2nd and 3rd degree A-V block (unless a permanent pacemaker is implanted)
* - severe bradycardia (heart rate <50)
* - 2nd and 3rd degree A-V block (unless a permanent pacemaker is implanted)
* - severe bradycardia (heart rate <50)
* - cardiogenic shock
* - sinus node dysfunction syndrome (including sinoatrial block)
* - severe hypotension (systolic blood pressure <85 mmHg)
* - Prinzmetal angina
* - untreated pheochromocytoma
* - metabolic acidosis
* - severe peripheral arterial circulation disorders
* - concurrent intravenous treatment with verapamil or diltiazem
* Additional exclusion criteria for patients using Spironolactone:
* - anuria
* - acute renal failure
* - severe renal impairment (estimated glomerular filtration rate <10 ml/min)
* - hyperkalemia >5.5 mmol/l
* - hyponatremia <125 mmol/l
* - Addison's disease
* - concurrent use of eplerenone or other potassium-sparing diuretics
* - porphyria
* Additional exclusion criteria for patients using Sacubitril/Valsartan:
* - concomitant use with Angiotensin converting enzyme (ACE) inhibitors
* - angioedema related to previous ACE inhibitor treatment or a history of angiotensin II receptor blockers (ARB) treatment
* - hereditary or idiopathic angioedema
* - concomitant use with medicinal products containing Aliskiren in patients with diabetes mellitus or in patients with impaired renal function (eGFR <60 ml/min/1.73 m2)
* - severe liver dysfunction, biliary cirrhosis and cholestasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Determination of the rate of significance between the serum concentration of the used medicinal products and the dose of this medicinal product | 24 month
  Determination whether the serum concentration of used medicinal products (Nebivolol, Valsartan/Sacubitril, Carvedilol, Bisoprolol, Metoprolol, Spironolactone) is more important than the dose of these medicinal products for compensating health status in patients with chronic heart failure with reduced ejection fraction (HFrEF).

SECONDARY OUTCOMES:
Clinical indicator - NT-proBNP concentration | 24 month
  Determination of a significant dependence between serum concentration of the used medicinal products and the values of the selected clinical indicator - N-terminal prohormone of natriuretic peptide B (NT-pro BNP), measured in pg/ml.
Clinical indicator - 6-minute walk test | 24 month
  Determination of a significant dependence between the serum concentration of the used medicinal products and the values of the selected clinical indicator - 6-minute walking test. The test measures the distance the patient walks 6 minutes in the corridor (in meters).
Clinical indicator - Minnesota Living With Heart Failure Questionnaire | 24 month
  Determination of a significant dependence between the serum concentration of the used medicinal products and the values of the selected clinical indicator - Minnesota Living With Heart Failure Questionnaire. The total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
Clinical indicator - Echocardiographic examination | 24 month
  Determination of a significant dependence between the serum concentration of the used medicinal products and the values of the selected clinical indicator - echocardiographic examination.
Clinical indicator - The hospitalization for HFrEF | 24 month
  Determination of a significant dependence between the serum concentration of the used medicinal products and the values of the selected clinical indicator - the hospitalization for HFrEF (yes/no).
Clinical indicator - The length of survival | 24 month
  Determination of a significant dependence between the serum concentration of the used medicinal products and the values of the selected clinical indicator - the length of survival (measured in month).
Adverse effects | 24 month
  Determination of the number of patients in whom a significant dependence between the serum concentration of the used medicinal products and the adverse effects of these medicinal products is demonstrated.
Non-adherence to treatment | 24 month
  Determination the number of patients in whom non-adherence to treatment will be demonstrated.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Lazárová, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Buda V, Prelipcean A, Cozma D, Man DE, Negres S, Scurtu A, Suciu M, Andor M, Danciu C, Crisan S, Dehelean CA, Petrescu L, Rachieru C. An Up-to-Date Article Regarding Particularities of Drug Treatment in Patients with Chronic Heart Failure. J Clin Med. 2022 Apr 4;11(7):2020. doi: 10.3390/jcm11072020. PMID 35407628
- [Background] Raschi E, Diemberger I, Sabatino M, Poluzzi E, De Ponti F, Potena L. Evaluating sacubitril/valsartan as a treatment option for heart failure with reduced ejection fraction and preserved ejection fraction. Expert Opin Pharmacother. 2022 Feb;23(3):303-320. doi: 10.1080/14656566.2022.2027909. Epub 2022 Jan 20. PMID 35050813
- [Background] Pyvovar SM, Rudyk IS. Use of beta-blockers in patients with heart failure - unresolved issues. Pol Merkur Lekarski. 2022 Aug 23;50(298):237-239. PMID 36086982
- [Background] Lee CM, Kang P, Cho CK, Park HJ, Lee YJ, Bae JW, Choi CI, Kim HS, Jang CG, Lee SY. Physiologically based pharmacokinetic modelling to predict the pharmacokinetics of metoprolol in different CYP2D6 genotypes. Arch Pharm Res. 2022 Jun;45(6):433-445. doi: 10.1007/s12272-022-01394-2. Epub 2022 Jun 28. PMID 35763157
- [Background] Fontana V, Turner RM, Francis B, Yin P, Putz B, Hiltunen TP, Ruotsalainen S, Kontula KK, Muller-Myhsok B, Pirmohamed M. Chromosomal Region 11p14.1 is Associated with Pharmacokinetics and Pharmacodynamics of Bisoprolol. Pharmgenomics Pers Med. 2022 Mar 22;15:249-260. doi: 10.2147/PGPM.S352719. eCollection 2022. PMID 35356681
- [Background] de Denus S, Leclair G, Dube MP, St-Jean I, Zada YF, Oussaid E, Jutras M, Givertz MM, Mentz RJ, Tang WHW, Ferreira JP, Rouleau J, Butler J, Kalogeropoulos AP. Spironolactone metabolite concentrations in decompensated heart failure: insights from the ATHENA-HF trial. Eur J Heart Fail. 2020 Aug;22(8):1451-1461. doi: 10.1002/ejhf.1802. Epub 2020 Apr 1. PMID 32237012
- [Background] Giri P, Joshi V, Giri S, Delvadia P, Jain MR. Simultaneous determination of sacubitrilat and fimasartan in rat plasma by a triple quad liquid chromatography-tandem mass spectrometry method utilizing electrospray ionization in positive mode. Biomed Chromatogr. 2021 Feb;35(2):e4981. doi: 10.1002/bmc.4981. Epub 2020 Sep 18. PMID 32895916
- [Background] Iacoviello M, Pugliese R, Correale M, Brunetti ND. Optimization of Drug Therapy for Heart Failure With Reduced Ejection Fraction Based on Gender. Curr Heart Fail Rep. 2022 Dec;19(6):467-475. doi: 10.1007/s11897-022-00583-w. Epub 2022 Oct 5. PMID 36197626
- [Background] Ritscher S, Georges C, Wunder C, Wallemacq P, Persu A, Toennes SW. Assessment of adherence to diuretics and beta-blockers by serum drug monitoring in comparison to urine analysis. Blood Press. 2020 Oct;29(5):291-298. doi: 10.1080/08037051.2020.1763775. Epub 2020 May 13. PMID 32400211
- [Background] Rea F, Iorio A, Barbati G, Bessi R, Castrichini M, Nuzzi V, Scagnetto A, Senni M, Corrao G, Sinagra G, Di Lenarda A. Patient adherence to drug treatment in a community based-sample of patients with chronic heart failure. Int J Cardiol. 2022 Feb 15;349:144-149. doi: 10.1016/j.ijcard.2021.11.018. Epub 2021 Nov 18. No abstract available. PMID 34801616
- [Background] Sweeney M, Cole GD, Pabari P, Hadjiphilippou S, Tayal U, Mayet J, Chapman N, Plymen CM. Urinary drug metabolite testing in chronic heart failure patients indicates high levels of adherence with life-prolonging therapies. ESC Heart Fail. 2021 Jun;8(3):2334-2337. doi: 10.1002/ehf2.13284. Epub 2021 Mar 11. PMID 33709563
- [Background] Simpson J, Jackson CE, Haig C, Jhund PS, Tomaszewski M, Gardner RS, Tsorlalis Y, Petrie MC, McMurray JJV, Squire IB, Gupta P. Adherence to prescribed medications in patients with heart failure: insights from liquid chromatography-tandem mass spectrometry-based urine analysis. Eur Heart J Cardiovasc Pharmacother. 2021 Jul 23;7(4):296-301. doi: 10.1093/ehjcvp/pvaa071. PMID 32597982
- [Background] Jelinek L, Vaclavik J, Ramik Z, Pavlu L, Benesova K, Jarkovsky J, Lazarova M, Janeckova H, Spurna J, Taborsky M. Directly Measured Adherence to Treatment in Chronic Heart Failure: LEVEL-CHF Registry. Am J Med Sci. 2021 Apr;361(4):491-498. doi: 10.1016/j.amjms.2020.12.004. Epub 2020 Dec 7. PMID 33781390